CLINICAL TRIAL: NCT01991912
Title: Irrigation Endoscopic Decompressive Laminotomy. A New Endoscopic Unilateral Approach for Bilateral Lumbar Decompression: A Blinded Non-randomized Controlled Trial.
Brief Title: Irrigation Endoscopic Decompressive Laminotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, hesham magdi soliman, doctor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IEDL
Record Dates: First submitted 2013-06-07; First posted 2013-11-25 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Lumbosacral Spinal Stenosis
Keywords: irrigation endoscopic decompression; minimally invasive surgery; spinal stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- irrigation endoscopic decompression (Experimental): endoscopic decompression is performed for cases of lumbar spinal stenosis.Portals 0.5cm in size are used for the introduction of the instruments and the endoscope. Saline under pump pressure is used to open a potential working space. This is followed by performing an ipsilateral hemilaminotomy and contralateral decompression under the midline structure
  Interventions: Procedure: open lumbar decompression

INTERVENTIONS:
Procedure: open lumbar decompression — A posterior midline incision is performed over the affected levels. Bilateral subperiosteal dissection of the paraspinal muscles is performed. Bilateral hemilaminotomies, foraminotomies and lateral recess decompression is performed followed by wound closure

SUMMARY:
The classic laminectomy for surgical treatment of spinal stenosis has considerable morbidity .This is further magnified by the disease being more common in elderly with associated medical comorbidities and being usually global involving multiple levels.The purpose of this study is to present and to evaluate a new endoscopic technique named Irrigation Endoscopic Decompressive Laminotomy (IEDL) for lumbar spinal canal decompression.

DETAILED DESCRIPTION:
In the IEDL group,2 portals 0.5cm were used one for the endoscope and the other for instruments. For every additional level one portal is added. The endoscope and instruments are directly placed over the surface of lamina without any dissection and saline under pump pressure is used to open a potential working space. Unilateral laminotomy and bilateral decompression under endoscopic vision is performed. In the microsurgical group, bilateral fenestration is performed in the usual manner

ELIGIBILITY:
Inclusion Criteria:

* neurogenic claudication,that correlated with moderate to severe spinal canal stenosis as shown on MRI and resistant to 3 months of conservative management .

Exclusion Criteria:

* predominant back pain or instability

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
oswestry disability index | 24 months

SECONDARY OUTCOMES:
postoperative hospital stay | 30 days
time required following surgery before return to work | 30 days
vas for back pain | 30 days

OTHER OUTCOMES:
complications | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: hesham m soliman, MD, Principal Investigator — Cairo University